CLINICAL TRIAL: NCT04195880
Title: Implementing and Evaluating INTERACT in VA CLCs
Brief Title: Reducing Veterans Hospitalizations From Community Living Centers
Acronym: INTERACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Providence VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CRE 12-025; CIRB 13-10 (Other: Providence VA Medical Center)
Record Dates: First submitted 2019-12-10; First posted 2019-12-12 (Actual); Results first posted 2020-05-11 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Quality Improvement

STUDY DESIGN:
Intervention Model Description: Pair matched cluster randomized trial; randomization at the provider level.
Masking Description: Intervention implemented in providers assigned to experimental condition, so all knew they were in a study. Control facilities did not know there was a study underway.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental VA Community Living Centers (Experimental): Eight VA CLCs selected to receive the INTERACT intervention
  Interventions: Other: Interventions to Reduce Acute Care Transfers
- Control VA Community Living Centers (No Intervention): Eight CLCs, matched to experiment CLCs, based on size, location to VAMC, and hospitalization rates, did not receive the intervention and continued care as usual

INTERVENTIONS:
Other: Interventions to Reduce Acute Care Transfers — Experimental CLCs were trained in INTERACT QI Intervention, containing tools, strategies and educational resources designed to catch and manage acute changes in conditions early that a Veteran may be experiencing, leading to a potential reduction in preventable hospital transfers from CLCs.
  Other Names: INTERACT
  Arms: Experimental VA Community Living Centers

SUMMARY:
The goal of the project was to implement and evaluate the intervention, Interventions to Reduce Acute Care Transfers (INTERACT) in VHA CLCs, which is designed to improve the care of Veterans using CLCs who experience acute changes in their condition and at the same time reduce their rate of hospitalization.

DETAILED DESCRIPTION:
The project was designed to show that engagement by frontline CLC staff, in using the INTERACT (VA version of INTERACT) program will identify Veterans' clinical problems earlier, help evaluate and safely initiate management of acute changes in conditions in the CLC, communicate more effectively with physicians about Veterans' conditions, thereby avoiding unnecessary hospitalizations, and provide more emergent hospitalizations when necessary.

The project planned to implement the INTERACT quality improvement program as the intervention in up to 15 randomly selected, pair matched CLCs for a 6 month intensive training period and an additional 12-18 month ongoing follow-up monitoring period.

Additionally, a quantitative and qualitative evaluation of the implementation of the INTERACT intervention was done to characterize the fidelity with which CLCs in the intervention pairs participated in training, engaged in regular conference calls, undertook root cause analyses identifying why hospitalizations occurred and used the tools in which they were trained.

The program's effect is based on three core strategies: 1) enabling front-line NH staff to identify acute conditions early in their course, thereby helping to prevent them from becoming severe enough to require acute hospitalization; 2) providing communication and decision support tools that assist with the safe and effective management of certain conditions in the Community Living Center (CLC) without transfer to the acute hospital; and 3) educating CLC staff in advance care planning and discussions about end-of-life and comfort care plans, and thus increasing the use of advance directives, comfort care measures, and palliative and hospice care as an alternative to hospitalization when appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Veterans in experimental and control CLCs during 18 months during which the INTERAC intervention was implemented.

Exclusion Criteria:

* Veterans not in participating CLCs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6543 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Mor, PhD, Principal Investigator — Providence VA Medical Center, Providence, RI
Locations (1):
- Providence VA Medical Center, Providence, RI, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mochel AL, Henry ND, Saliba D, Phibbs CS, Ouslander JG, Mor V. INTERACT in VA Community Living Centers (CLCs): Training and Implementation Strategies. Geriatr Nurs. 2018 Mar-Apr;39(2):212-218. doi: 10.1016/j.gerinurse.2017.09.002. Epub 2017 Oct 5. PMID 28988835
- [Result] Mochel AL, Holle CL, Rudolph JL, Ouslander JG, Saliba D, Mor V, Mittman BS. Influencing Factors Associated with Implementation of INTERACT (Interventions to Reduce Acute Care Transfers) in VA Community Living Centers (CLCs) Using the Consolidated Framework. J Aging Soc Policy. 2022 Sep 3;34(5):673-689. doi: 10.1080/08959420.2021.1926862. Epub 2021 Jun 4. PMID 34085597
- See also: Related Info — https://doi.org/10.1016/j.gerinurse.2017.09.002

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All Veterans admitted to any of the eight experimental and eight control facilities (VA Community Living Centers) during the study timeframe, January 2016 - December 2017.
Period: Overall Study
Arm/Group | Experimental VA Community Living Centers | Control VA Community Living Centers
Started | 3205 | 3338
Completed | 3205 | 3338
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental VA Community Living Centers | Control VA Community Living Centers | Total
Number analyzed (Participants) | 3205 | 3338 | 6543
Age, Customized [Count of Participants; unit: Participants]
  <55 | 121 | 141 | 262
  55-64 | 542 | 583 | 1125
  65-74 | 1187 | 1150 | 2337
  75-84 | 673 | 656 | 1329
  85+ | 682 | 808 | 1490
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 84 | 194
  Male | 3095 | 3254 | 6349
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, non-Hispanic | 2308 | 2374 | 4682
  Black | 788 | 816 | 1604
  Hispanic | 47 | 79 | 126
  Other | 28 | 39 | 67
  Unknown | 34 | 30 | 64
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3205 | 3338 | 6543

OUTCOME MEASURES:

1. Primary Outcome: Hospital Admissions Per Person Year Alive Measured at the Facility Month Level
Description: hospital admissions from nursing home per person year at risk of being hospitalized calculated for each of the 16 facilities per month of observation during the 18 months of the active study and 18 months preceding introduction of the intervention in the experimental facilities. This measure is constructed from EMR data and not from a scale.
Time Frame: 36 months
Measure: Mean (Standard Error); unit: hospitalizations per person year alive
Arm/Group | Experimental VA Community Living Centers | Control VA Community Living Centers
Number analyzed (Participants) | 3205 | 3338
hospitalizations per person year alive | 5.5 (2.5) | 5.8 (2.5)
Statistical Analysis 1: Comparison: Experimental VA Community Living Centers vs Control VA Community Living Centers; We assumed the average monthly pre-intervention hospitalization rates of intervention and control CLCs were equal, so only average monthly post-intervention hospitalization rates might diverge. Each CLC had its own start month and contributed 18 months pre-intervention and 18 months post-intervention. Hospitalizations rates were modeled using a multilevel negative-binomial regression because it allows for over-dispersion, which is commonly observed with medical events such as a count; Test type: Superiority; p < .05, negative-binomial regression coefficient

2. Secondary Outcome: Potentially Avoidable Hospitalizations
Description: Potentially avoidable hospitalization per person year alive aggregated to the facility level. These hospitalizations are a sub-set of all hospitalizations based upon an AHRQ algorithm frequently referenced in the literature.
Time Frame: 18 months followup during observation period.
Measure: Number (95% Confidence Interval); unit: hospitalizations per person year alive
Arm/Group | Experimental VA Community Living Centers | Control VA Community Living Centers
Number analyzed (Participants) | 3205 | 3338
hospitalizations per person year alive | .3 [0.0 to 1.4] | .2 [0 to 1.3]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the study timeframe (18 Months, introduction of intervention, implementation and monitoring) for the eight experimental CLC Veterans and eight controls
Description: To ensure the safety of Veterans in the CLC and confirm the intervention is not reducing hospitalizations to the detriment of Veterans', we had a safety monitoring plan in place which was reviewed and signed off by the Data Safety Monitoring Board (DSMB) and we generated mortality data for all CLC residents in both INTERACT (experimental) and control facilities, charting changes in mortality rates relative to the historical and contemporary mortality rates of paired facilities.
Arm/Group | Experimental VA Community Living Centers | Control VA Community Living Centers
All-Cause Mortality (participants affected / at risk) | 0/3205 | 0/3338
Serious Adverse Events (participants affected / at risk) | 0/3205 | 0/3338
Other Adverse Events (participants affected / at risk) | 0/3205 | 0/3338

LIMITATIONS AND CAVEATS:
Our intervention and control CLCs were not perfectly matched. Due to incomplete implementation of INTERACT in all intervention sites, we acknowledge that this was an incomplete test of the efficacy of the program when properly implemented

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-28): https://cdn.clinicaltrials.gov/large-docs/80/NCT04195880/Prot_SAP_000.pdf